CLINICAL TRIAL: NCT05308082
Title: Programme Evaluation on Effectiveness of The Use of Movement-based x 'Elderspirituality - Fu Le Mun Sum' Intervention to Support Elderly People With Depressive Symptoms
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Collaborators: Tung Wah Group of Hospitals (Other)
Responsible Party: Principal Investigator, Prof. Vivian W.Q. Lou, Associate Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: RS200375
Record Dates: First submitted 2022-03-24; First posted 2022-04-01 (Actual); Last update posted 2023-05-09 (Actual); Status verified 2023-05

CONDITIONS: Depression in Old Age
Keywords: Depression; Dance Movement Therapy; Depressive symptoms; Older adults; Elderly; Ageing
MeSH Terms: conditions — Depression

STUDY DESIGN:
Intervention Model Description: It is proposed that a total of 140 participants will be recruited, with 70 assigned to the intervention group, and 70 to the active control group. For the active control group, health talk will be delivered to participants which will match the length of contact and interval of contact of that in the intervention group. For the intervention group, dance movement therapy will be delivered on a regular basis.
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Experimental): It is proposed to have 70 participants who meet the inclusion criteria in the intervention group. Dance movement therapy will be delivered as an intervention, which consists of six sessions: (1) Movement for Self-expression, (2) Movement for Emotional Health I, (3) Movement for Emotional Health II, (4) Movement for Connection & Creativity, (5) Embracing your Dancing Child, and (6) Movement for Self-compassion.
  Interventions: Behavioral: Dance Movement Therapy (DMT)
- Active control group (No Intervention): It is proposed to have 70 participants who meet the inclusion criteria in the active control group. Health talk will be delivered to participants which will match the length of contact and interval of contact of that in the intervention group.

INTERVENTIONS:
Behavioral: Dance Movement Therapy (DMT) — The main Dance Movement Therapy (DMT) methods were dance-movement improvisations, body awareness exercises, and reflection through drawing/painting, writing, and verbalization. There was an orientation to personal space and body awareness, interaction in pairs, and interaction in the whole group. The themes included exploration of boundaries, somatic resources, symbols, pleasant and unpleasant emotions, mindfulness, and body awareness, enriched movement experiences, and safety and touch. In the present study, it consists of six sessions, including (1) Movement for Self-expression, (2) Movement for Emotional Health I, (3) Movement for Emotional Health II, (4) Movement for Connection & Creativity, (5) Embracing your Dancing Child, and (6) Movement for Self-compassion.
  Arms: Intervention group

SUMMARY:
Depression is one of the most common mood disorders in old age, and yet it is frequently under-detected and under-treated. Adopting a train-the-trainer approach, this project intends to utilize the dance movement therapy (DMT), as intervention, to support elderly people with depressive symptoms.

DETAILED DESCRIPTION:
In the present project, two evaluation studies will be conducted. The first study will evaluate the effectiveness of a train-the-trainer approach provided to frontline art development officers who will subsequently conduct interventions for the elderly. A participatory train-the-trainer approach will be adopted to develop a new intervention protocol by integrating body-movement therapeutic elements and a spiritual well-being enhancement group. In the second study, a quasi-experimental design will be adopted to examine the effectiveness of the Movement-based x 'Elderspirituality - Fu Le Mun Sum' intervention to support elderly people with depressive symptoms.

ELIGIBILITY:
Inclusion Criteria:

* aged 60 or above
* physical mobility of at least the limbs and body
* sufficient visual and auditory abilities to complete assessments
* with a clinical diagnosis of depression or with depressive symptoms (measured as the sum of 4 dichotomous items of the Geriatric Depression Scale)

Exclusion Criteria:

- a clinical diagnosis of severe illness that led to neurological deficits which limits the participation during the intervention

Ages: 60 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 135 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2022-12-24 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
Spirituality Scale for Chinese Elders (SSCE) | 4 months
  SSCE is a self-rated instrument that consists of 44 items to assess spiritual well-being among Chinese elders, covering 8 core elements: (1) meaning of life, (2) spiritual well-being, (3) transcendence, (4) relationship with self, (5) relationship with family, (6) relationship with others (friends and people around you), (7) relationship with the environment, and (8) relationship with life and death. Responses are rated on a 5-point Likert scale with scores ranging from 0 (never) to 4 (always) to measure the frequency of a certain perception or behaviour.

SECONDARY OUTCOMES:
The 15-item Geriatric Depression Scale (GDS-15) | 4 months
  It is a widely used screening instrument for depressive symptoms in the elderly. It consists of 15 items on a checklist; the response to each statement is either "yes" or "no".
The 5-level EQ-5D version (EQ-5D-5L) | 4 months
  This is a valid and widely used scale with 6 items to measure the quality of life among the general population. The EQ-5D-5L essentially consists of 2 facets: the EQ-5D descriptive system and the EQ visual analogue scale (EQ-VAS). The descriptive system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, several problems, and extreme problems. The EQ-VAS records the patient's self-rated health on a vertical visual analogue scale, where the endpoints are labelled "The best health you can imagine" and "The worst health you can imagine"

CONTACTS AND LOCATIONS:
Overall Officials: Vivian W. Q. Lou, PhD, Principal Investigator — The University of Hong Kong
Locations (1):
- Sau Po Centre on Ageing, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Data collected in this study will be published and submitted to academic journals and as research report to share with other researchers and practitioners.
Supporting Information: Study Protocol, CSR
Time Frame: No limitations on the publications
Access Criteria: No limitations on the publications